CLINICAL TRIAL: NCT02028364
Title: Pet Imaging as a Biomarker of Everolimus Added Value in Hormone Refractory postmenopausaL Women
Brief Title: Pet Imaging as a Biomarker in Hormone Refractory postmenopausaL Women
Acronym: PEARL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-BCTL:20120306; 2012-004860-22 (EudraCT Number)
Record Dates: First submitted 2013-11-20; First posted 2014-01-07 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Locally advanced breast cancer; HER2 negative; NSAI refractory; Metastatic breast cancer; Estrogen-receptor positive (ER+)
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus given in conjunction with exemestane (Experimental): Everolimus 10mg orally daily given in conjunction with exemestane 25mg orally daily until disease progression or treatment discontinuation for any other reasons.
  Interventions: Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Everolimus — 10mg orally daily
  Other Names: Afinitor
Drug: Exemestane — 25mg orally daily
  Other Names: Aromasin, Exemestane Teva, Exemestane Sandoz, Exemarom,Exemestane Mylan, Exemestane Accord Healthcare

SUMMARY:
This is a prospective, single arm trial in which patients with locally advanced or metastatic endocrine receptor positive and HER2 negative breast cancer refractory to non-steroidal aromatase inhibitors (NSAI) will receive Everolimus 10mg orally daily given in conjunction with exemestane 25mg orally daily until disease progression or treatment discontinuation for any other reasons. The main objectives are to evaluate if early metabolic response (MR) using FDG-PET/CT is associated with progression free survival (PFS) and overall survival (OS) in this population.

Tumour, metastatic lesions and blood samples will be collected during the treatment period in order to identify biomarkers predicting resistance to study treatment. Results will be correlated with the results of early FDG PET/CT data in order to better characterise the non-responders.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥18 years of age) with locally advanced or metastatic breast cancer not amenable to curative treatment by surgery or radiotherapy.
2. Histological or cytological confirmation of estrogen-receptor positive (ER+), HER2 negative breast cancer.
3. Postmenopausal female defined as:

   * Age ≥55 years and one year or more of amenorrhoea
   * Age <55 years and one year or more of amenorrhoea, with an estradiol assay <20pg/ml
   * Surgical menopause with bilateral oophorectomy NOTE: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LHRH) agonist (goserelin or leuprolide) is not permitted for induction of ovarian suppression.
4. Breast cancer that is refractory to non-steroidal aromatase inhibitors (NSAI) (i.e. anastrozole or letrozole) defined as:

   * Recurrence while on, or within 12 months of end of adjuvant treatment with anastrozole or letrozole; OR
   * Progression while on, or within one month of end of anastrozole or letrozole or treatment for locally advanced or metastatic breast cancer.

   NOTE: Letrozole or anastrozole do not have to be the last treatment prior to enrolment.
5. FDG-PET measurable disease defined as: at least one target lesion fulfilling following criteria:

   * Size ≥1.5cm; AND
   * FDG-PET avid lesion with uptake above the background liver uptake as described below: i.e. with a marked accumulation of FDG, at least 1.5-fold greater than liver SUV mean + 2 SDs (in 3cm spherical ROI in normal right lobe of liver). If liver is abnormal, target lesion should have uptake > 2.0 x SUV mean of blood pool in 1cm diameter ROI in descending thoracic aorta)

   NB:
   * The target lesion can be a bone metastasis if it fulfils the above mentioned criteria.
   * In the case the target lesion is a lymph node, the small axis should be ≥ 1.5cm.
6. Radiological or clinical evidence of recurrence or progression on last systemic therapy prior to enrolment.
7. Adequate bone marrow function as shown by:

   * Haemoglobin (HgB) ≥9.0 g/dL
   * ANC ≥1,500/mm3 (≥1.5 x 109/L)
   * Platelets ≥100,000/mm3 (≥100x 109/L)
8. Adequate liver function as shown by:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5xULN (or ≤5 if hepatic metastases are present)
   * Total serum bilirubin ≤1.5 x ULN (≤3 ULN for patients known to have Gilbert Syndrome)
9. Adequate renal function as shown by Serum creatinine ≤1.5 x ULN
10. Fasting serum cholesterol, triglycerides and glucose

    * Fasting serum cholesterol ≤300 mg/dL or 7.75 mmol/L
    * Fasting triglycerides ≤2.5 x ULN
    * Fasting glucose < 1.5 x ULN
11. Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2.
12. Written and signed informed consent obtained before any trial related activity.
13. Availability of a FFPE core of primary breast tumor
14. Possibility to obtain the mandatory blood samples for the translational research studies.
15. For patients with accessible metastatic lesions, possibility to obtain the mandatory biopsy (FFPE and frozen) of a metastatic lesion

Exclusion criteria:

1. HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
2. Patients with only non-measurable lesions by FDG-PET/CT (e.g. pleural effusion, ascites etc.).
3. Symptomatic visceral disease for example liver, pulmonary metastases or lymphangitis carcinomatosis.
4. Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin).
5. Another malignancy within 5 years prior to enrolment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer.
6. Radiotherapy within four weeks prior to enrolment except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture, which can then be completed within two weeks prior to enrolment. Patients must have recovered from radiotherapy toxicities prior to enrolment.
7. Currently receiving hormone replacement therapy, unless discontinued prior to enrolment.
8. Symptomatic brain metastases or other central nervous system metastases which are not controlled by local treatments.
9. Patients receiving concomitant immunosuppressive agents or chronic corticosteroid use at the time of study entry except in cases outlined below:

   * Topical applications (e.g. rash)
   * Inhaled sprays (e.g. obstructive airways disease)
   * Eye drops
   * Local injections (e.g. intra-articular)
   * Stable low dose of corticosteroids for at least two weeks before enrolment
10. Patients with known HIV seropositivity. Screening for HIV infection at baseline is not required
11. Acute and chronic, active infectious disorders (except for Hepatitis B and Hepatitis C positive patients).
12. Active bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin, LMWH and acetylsalicylic acid or equivalent, as long as the INR is ≤ 2.0).
13. Any severe uncontrolled medical conditions such as:

    * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to enrolment, uncontrolled cardiac arrhythmia
    * Uncontrolled diabetes as defined by fasting glucose ≥ 1.5 x ULN
    * Acute and chronic, active infectious disorders and non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy.
    * Symptomatic deterioration of lung function
14. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazoleonazole, Voriconazole, Ritonavir, Telithromycin) within the last 5 days prior to enrolment.
15. History of non-compliance to medical regimens.
16. Patients unwilling or unable to comply with the protocol.
17. Concurrent anti-cancer treatment in another investigational trial, including hormonal therapy, immunotherapy or targeted agents other than those administered in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01-12; Primary Completion 2021-07-06 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
PFS based on RECIST criteria 1.1. | 2.5 years from FPI
  To evaluate if early metabolic response (MR) using FDG-PET/CT is associated with progression free survival (PFS) in ER+, HER2 negative ABC or MBC patients treated with exemestane plus everolimus.

SECONDARY OUTCOMES:
Overall survival (OS) | 2.5 years from first patient in
  To evaluate if early metabolic response (MR) using FDG-PET/CT is associated with overall survival (OS) in ER+, HER2 negative locally advanced or MBC patients treated with exemestane plus everolimus.
* Proportion of FDG-PET/CT metabolic non-responders/FDG-PET/CT metabolic responders * Estimate the most suitable second FDG-PET/CT time point (2 weeks versus 4 weeks after initiation of treatment). | Baseline, day 14, Day 28 and at progression
  FDG PET/CT will be done three times during the pilot phase of the study (first 30 patients): at baseline (at day 0, Day 14 and day 28). FDG PET/CT will be done twice during the extension phase: at baseline (at day 0, Day 14 or Day 28) depending the results of the pilot phase.
Biomarker Assessment | baseline, day 14, day 28, every 12 weeks and at progression
  The aim is to identify biomarkers predicting resistance to exemestane and everolimus therapy by studying primary tumor, metastatic biopsies and serial plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gombos, MD, Principal Investigator — Insitut Jules Bordet; Patrick Flamen, MD, Principal Investigator — Jules Bordet Institute
Locations (5):
- Belgium (5):
  - institut Jules Bordet, Brussels
  - Cliniques Universtaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - CHU Ambroise Paré, Mons
  - Clinique et Maternité Sainte Elisabeth, Namur